CLINICAL TRIAL: NCT00513747
Title: A Phase III Intergroup CLL Study of Asymptomatic Patients With Untreated Chronic Lymphocytic Leukemia Randomized to Early Intervention Versus Observation With Later Treatment in the High Risk Genetic Subset With IGVH Unmutated Disease
Brief Title: Early or Delayed Fludarabine and Rituximab in Treating Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-10501; U10CA031946 (NIH); CDR0000537685 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive rituximab IV over 4 hours on days 1, 3, and 5 of week 1 and then on day 1 of weeks 5, 9, 13, 17, and 21. Patients also receive fludarabine phosphate IV over 30 minutes on days 1-5 of weeks 1, 5, 9, 13, 17, and 21. After completion of chemoimmunotherapy, patients are followed every 3 months until disease progression. At the time of disease progression, patients receive retreatment with chemoimmunotherapy as above or another treatment regimen.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate
- Arm II (Active Comparator): Patients are followed every 3 months until disease progression. At the time of disease progression, patients receive rituximab and fludarabine phosphate as in arm I. Patients are then followed every 3 months until second disease progression. Patients with a second disease progression receive retreatment with chemoimmunotherapy as above or another treatment regimen.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: rituximab — Given IV over 4 hours
Drug: fludarabine phosphate — Given IV over 30 minutes

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving fludarabine together with rituximab may kill more cancer cells. Sometimes the cancer may not need treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether giving fludarabine together with rituximab early is more effective than giving fludarabine and rituximab after observation in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying fludarabine and rituximab to compare how well they work when given early or after observation in treating patients with previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if early treatment with chemoimmunotherapy comprising fludarabine phosphate and rituximab extends the time to second treatment in patients with genetically high-risk (unmutated IgV_H), asymptomatic, previously untreated chronic lymphocytic leukemia (CLL).
* To determine the time to disease progression that would warrant second treatment.
* To determine overall survival.

Secondary

* To measure the proportion of patients with asymptomatic, previously untreated CLL who have mutated and unmutated IgV_H genes.
* To determine the differences in acute and chronic toxicity of administering chemoimmunotherapy early to patients with genetically high-risk CLL compared to waiting until symptoms develop.
* To determine the effect of select pretreatment clinical and biological characteristics (such as interphase cytogenetic abnormalities, ZAP-70 expression, and p53 dysfunction [primary and secondary]) on response, time to second treatment, and overall survival of patients with genetically high-risk CLL randomized to early treatment.
* To determine the effect of select pretreatment clinical and biological characteristics (such as interphase cytogenetic abnormalities, ZAP-70 expression, and p53 dysfunction) on response, time to first and second treatments, and overall survival of patients with genetically high-risk CLL randomized to standard treatment (observation until symptoms occur).
* To describe the natural history of patients with genetically low-risk (mutated IgV_H genes), asymptomatic, previously untreated CLL, in terms of time to initial treatment, response, progression, and survival.
* To determine the effect of select pretreatment characteristics on time to first treatment, response, progression, and survival of patients with genetically low-risk CLL.
* To correlate patterns of resistance that emerge in patients with unmutated IgV_H genes who have relapsing or refractory CLL following receipt of chemoimmunotherapy with clonal evolution, including acquisition of high-risk karyotype abnormalities, p53 mutations, p53 dysfunction (primary and secondary), altered mRNA and protein expression related to treatment resistance, DNA mutations, microRNA gene expression, and methylation changes.
* To determine whether highly sensitive flow cytometry negativity at completion of therapy in patients randomized to early treatment is an effective surrogate marker for prolonged time to second treatment, overall survival, and other clinical benefits.
* To collect demographic data on familial CLL in newly diagnosed patients participating on this study.

OUTLINE: This is a multicenter study.

* Genetically high-risk disease: Patients are stratified according to age (< 50 years vs 50 to 70 years vs > 70 years) and presence of the high-risk genetic feature [del(11)(q22.3) or del(17)(p13.1)] by FISH (yes vs no). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive rituximab IV over 4 hours on days 1, 3, and 5 of week 1 and then on day 1 of weeks 5, 9, 13, 17, and 21. Patients also receive fludarabine phosphate IV over 30 minutes on days 1-5 of weeks 1, 5, 9, 13, 17, and 21. After completion of chemoimmunotherapy, patients are followed every 3 months until disease progression. At the time of disease progression, patients receive retreatment with chemoimmunotherapy as above or another treatment regimen.
  * Arm II: Patients are followed every 3 months until disease progression. At the time of disease progression, patients receive rituximab and fludarabine phosphate as in arm I. Patients are then followed every 3 months until second disease progression. Patients with a second disease progression receive retreatment with chemoimmunotherapy as above or another treatment regimen.
* Genetically low-risk disease: Patients are followed every 3 months until disease progression. At the time of disease progression, patients receive rituximab and fludarabine phosphate as in arm I. Patients are then followed every 3 months until second disease progression. Patients with a second disease progression receive retreatment with chemoimmunotherapy as above or another treatment regimen.

Patients undergo blood sample collection periodically for correlative studies.

After finishing treatment, patients are followed periodically.

ELIGIBILITY:
Eligibility Criteria for Pre-Registration:

1. Patients must be within 6 months of the initial flow cytometric confirmation of B-cell chronic lymphocytic leukemia (CLL). This interval begins with the initial flow cytometric confirmation of disease.
2. Clinical and immunophenotypic evidence of CLL including:

   2.1 An absolute lymphocytosis of > 5,000/μL
   * Morphologically, the lymphocytes must appear mature with < 55% prolymphocytes.
   * Local institution lymphocyte phenotype must reveal a predominant B-cell monoclonal population sharing a B-cell marker (CD19, CD20, CD23) with the CD5 antigen, in the absence of other pan-T-cell markers.
   * Additionally, the B-cells must be monoclonal with regard to expression of either κ or λ and have surface immunoglobulin expression of low density.
   * Patients with bright surface immunoglobulin levels must have CD23 coexpression and absence of t(11;14) on interphase cytogenetics or have negative tumor protein staining for cyclin D1.

   2.2 Staging - Patients must be in the low category (i.e., only stages 0 or I) of the modified three-stage Rai staging system as described in the protocol.
3. Patients should not have evidence of active disease as demonstrated by any of the following criteria:

   * Splenomegaly and/or massive/progressive lymphadenopathy that would require therapy
   * Presence of weight loss > 10% over the preceding 6 month period
   * Grade 2 or 3 fatigue
   * Fevers > 100.5°F or night sweats for greater than 2 weeks without evidence of infection
   * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of less than 6 months.
4. Prior Treatment: No prior therapy for CLL including corticosteroids for autoimmune complications that have developed since the initial diagnosis of CLL.
5. Age ≥ 18 years
6. Performance Status 0 - 1.
7. No HIV disease. Due to alterations in host immunity, patients known to have HIV infection may not be enrolled.
8. Non-pregnant and non-nursing. Due to the unknown teratogenic potential of chemotherapy, pregnant or nursing women may not be enrolled. Women and men of reproductive potential should agree to use an effective means of birth control.
9. Required Initial Laboratory Values:

   * Creatinine ≤ 1.5 x upper limit of normal

Eligibility Criteria for Registration (to Low-Risk Cohort or High-Risk Cohort Randomization between Early Intervention Versus Observation with Later Treatment)

1. Successful determination of IgVH mutational status by reference laboratory.
2. Absence of progression of CLL, i.e., absence of the following:

   * Progressive splenomegaly and/or lymphadenopathy on two independent measures spaced two weeks apart. If one assessment notes progression, this should be repeated prior to re-registration.
   * Development of anemia (hemoglobin < 11 g/dL) or thrombocytopenia (platelets < 100,000/μL).
   * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of less than 6 months.
   * Symptoms referable to CLL, including weight loss > 10% over the preceding 6 month period; grade 2 or 3 fatigue; or fevers > 100.5°F and/or night sweats for greater than 2 weeks without evidence of infection.
3. Required Laboratory Value:

   * Creatinine ≤ 1.5 x upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Byrd, MD, Study Chair — Ohio State University
Locations (387):
- United States (379):
  - Regional Medical Center, Anniston, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Memorial Medical Center, Modesto, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Central Dupage Cancer Center, Winfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - MaineGeneral Medical Center - Waterville, Waterville, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (8):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Derived] Deshields TL, Dueck AC, Rogers K, Brown JR, Shanafelt T, Mintzer D, Byrd JC. Perceived risk for cancer progression and psychological status in chronic lymphocytic leukemia patients: CALGB 70603 (Alliance). Leuk Lymphoma. 2019 Oct;60(10):2580-2583. doi: 10.1080/10428194.2019.1594218. Epub 2019 Mar 27. PMID 30916608

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Enrollment number in the Protocol Section does not match the number of participants who started in the Participant Flow due to limited data on one participant (i.e. the participant was registered but was not randomized or classified (high vs. low risk) because the participant withdrew consent for all follow-up the same day of registration).
Groups:
- Arm A: High Risk Early Intervention: Randomized Patients receive 50, 325, and 375 mg/m^2 rituximab IV over 4 hours on days 1, 3, and 5 of week 1, respectively; then patients receive 375 mg/m^2 rituximab IV on day 1 of weeks 5, 9, 13,
  > 17, and 21. Patients also receive 25 mg/m^2/day fludarabine monophosphate IV over 30 minutes on days 1-5 of weeks 1, 5, 9, 13, 17, and 21. After completion of chemoimmunotherapy, patients are followed every 3 months until disease progression. At the time of disease progression, patients receive retreatment with chemoimmunotherapy as above or another treatment regimen.
- Arm B: High Risk Observation + Later Treatment: Randomized Patients are followed every 3 months until disease progression. At the time of disease progression, patients receive rituximab and fludarabine phosphate as in Arm A. Patients are then followed every 3 months until second disease progression. Patients with a second disease progression receive retreatment with chemoimmunotherapy as above or another treatment regimen.
- Arm C: Low Risk Observation + Later Treatment: Patients who were registered to the low-risk arm may elect to provide continued follow-up information on their treatment, disease course, and outcome regardless of the medical therapy they and their physician select. Patients are followed every 3 months until disease progression. At the time of disease progression, patients receive rituximab and fludarabine phosphate as in Arm A. Patients are then followed every 3 months until second disease progression. Patients with a second disease progression receive retreatment with chemoimmunotherapy as above or another treatment regimen.
Period: Overall Study
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment | Arm C: Low Risk Observation + Later Treatment
Started | 17 | 11 | 55
Received at Least One Dose of Treatment (Participants received at least one dose of treatment and were evaluated for adverse events.) | 9 | 11 | 40
Completed | 17 | 11 | 55
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: High Risk Early Intervention: Randomized Patients receive 50, 325, and 375 mg/m^2 rituximab IV over 4 hours on days 1, 3, and 5 of week 1, respectively; then patients receive 375 mg/m^2 rituximab IV on day 1 of weeks 5, 9, 13,> 17, and 21. Patients also receive 25 mg/m^2/day fludarabine monophosphate IV over 30 minutes on days 1-5 of weeks 1, 5, 9, 13, 17, and 21. After completion of chemoimmunotherapy, patients are followed every 3 months until disease progression. At the time of disease progression, patients receive retreatment with chemoimmunotherapy as above or another treatment regimen.
- Total: Total of all reporting groups
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment | Arm C: Low Risk Observation + Later Treatment | Total
Number analyzed (Participants) | 17 | 11 | 55 | 83
Age, Continuous [Median (Full Range); unit: years] | 60 [45 to 80] | 60 [49 to 76] | 59 [39 to 81] | 60 [39 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 23 | 27
  Male | 16 | 8 | 32 | 56

OUTCOME MEASURES:

1. Primary Outcome: Time to Second Treatment in High Risk Patients
Description: Kaplan-Meier analysis was conducted to estimate the distribution of time from randomization to second treatment or death whichever comes first. Events were defined as the start of second treatment or death. Patients who had not experienced one of these defined events of interest were censored at their last known follow-up.
Time Frame: Up to 72 months
Population: Randomized High Risk patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment
Number analyzed (Participants) | 17 | 11
months | 62.7 [57.3 to 66.5] | 56.3 [39.2 to 56.3]
Statistical Analysis 1: Comparison: Arm A: High Risk Early Intervention vs Arm B: High Risk Observation + Later Treatment; Test type: Superiority; p = 0.1521, Log Rank

2. Primary Outcome: Disease-Free Survival in High Risk Patients
Description: Kaplan-Meier analysis was conducted to estimate disease free survival defined as:>
  * Arm A: Time from randomization until Second Treatment (first relapse) or death whichever comes first. Events were defined as the start of second treatment or death. Patients who had not experienced one of these defined events of interest were censored at their last known follow-up.>
  * Arm B: Time from randomization until First Treatment (first relapse) or death whichever comes first. Events were defined as the start of first treatment or death. Patients who had not experienced one of these defined events of interest were censored at their last known follow-up.
Time Frame: Up to 72 months
Population: Randomized High Risk patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment
Number analyzed (Participants) | 17 | 11
months | 62.7 [57.3 to 66.5] | 39.2 [33.9 to NA] — The 95% confidence interval upper limit was not evaluable (i.e. under the level of detection).
Statistical Analysis 1: Comparison: Arm A: High Risk Early Intervention vs Arm B: High Risk Observation + Later Treatment; Test type: Superiority; p = 0.0097, Log Rank

3. Primary Outcome: Overall Survival (OS) for High Risk Patients
Description: Kaplan-Meier analysis was conducted to estimate the distribution of time from randomization to death from any cause. Estimates were not stratified. Patients who did not experience this primary outcome had their survival times censored at their last follow-up.
Time Frame: Up to 72 months
Population: Randomized High Risk patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment
Number analyzed (Participants) | 17 | 11
months | NA [NA to NA] — The median and 95% confidence interval are not evaluable (i.e. under the level of detection). | NA [39.2 to NA] — The median and 95% confidence interval upper limit are not evaluable (i.e. under the level of detection).
Statistical Analysis 1: Comparison: Arm A: High Risk Early Intervention vs Arm B: High Risk Observation + Later Treatment; Test type: Superiority; p = 0.4645, Log Rank

4. Secondary Outcome: Number of Patients With Mutated and Unmutated IgVH Genes
Description: Number of patients with mutated and unmutated IgVH genes are reported below.
Time Frame: Once at baseline
Population: All patients are included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Arm A + Arm B + Arm C patients
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment | Arm C: Low Risk Observation + Later Treatment | Total
Number analyzed (Participants) | 17 | 11 | 55 | 83
Participants
  Unmutated | 17 | 11 | 0 | 28
  Mutated | 0 | 0 | 55 | 55

5. Secondary Outcome: Overall Survival in Low Risk Patients
Description: Overall survival in low risk patients (registration to first treatment or death)>
  • Events were defined as death from any cause. Low risk Patients who were alive were censored at their last known follow-up.
Time Frame: Up to 72 months
Population: Low Risk patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C: Low Risk Observation + Later Treatment
Number analyzed (Participants) | 55
months | 58.1 [58.1 to NA] — The 95% confidence interval upper limit was not evaluable (i.e. under the level of detection).

6. Secondary Outcome: Time to First Treatment Survival in Low Risk Patients
Description: Time to First Treatment Survival in low risk patients (registration to first treatment or death)>
  • Events were defined as the start of first treatment or death from any cause. Patients who didn't receive their first treatment were censored at their last known follow-up.
Time Frame: Up to 72 months
Population: Low Risk patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C: Low Risk Observation + Later Treatment
Number analyzed (Participants) | 55
months | 58.1 [58.1 to 70.3]

ADVERSE EVENTS:
Time Frame: Up to 72 months
Description: Participants who received at least one dose of treatment are evaluable for adverse events (AEs) (i.e. summarized in the Serious and Other(Not Including Serious) AEs tables). All participants are followed for their survival status (i.e. summarized in the All-Cause Mortality table).
Arm/Group | Arm A: High Risk Early Intervention | Arm B: High Risk Observation + Later Treatment | Arm C: Low Risk Observation + Later Treatment
All-Cause Mortality (participants affected / at risk) | 1/17 | 2/11 | 2/55
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/40
Other Adverse Events (participants affected / at risk) | 9/9 | 11/11 | 40/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: High Risk Early Intervention (N=9) | Arm B: High Risk Observation + Later Treatment (N=11) | Arm C: Low Risk Observation + Later Treatment (N=40)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (25) | 5 (16) | 16 (43)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (8) | 1 (1) | 2 (3)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (32) | 9 (30) | 19 (70)
General symptom (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastric infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingival infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious meningitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lip infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa(unknown ANC) (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Pharyngitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Rhinitis infective(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 6 (7)
Sinusitis(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 7 (7)
Ureteritis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (3) | 1 (6)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 4 (6) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (16) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (21) | 2 (5) | 8 (22)
Platelet count decreased (Investigations) | 5 (21) | 4 (17) | 14 (55)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Weight gain (Investigations) | 1 (3) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (11)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (14)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (2) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (3) | 2 (4)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (4)
Depression (Psychiatric disorders) | 1 (1) | 4 (24) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (3) | 2 (5) | 2 (2)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 5 (14) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (6) | 2 (6) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (2)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 2 (4)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes